CLINICAL TRIAL: NCT05511064
Title: A Multiple Center, Clinical Trial to Evaluate the Efficacy and Safety of Blood Circulation Improvement Using an Investigational Device (Model Name CGM MB-1701) for the Risk Group of Deep Vein Thrombosis (DVT)
Brief Title: CEFID-II (CEra Flow Improves DVT-II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ceragem Clinical Inc. (Industry)
Responsible Party: Sponsor
Organization: Ceragem Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CGM-21-031
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Blood Circulation Disorder; Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- blood circulation treatment (Experimental): Blood circulation treatment for the risk group for Deep Vein Thrombosis (DVT)
  Interventions: Device: Blood circulation device

INTERVENTIONS:
Device: Blood circulation device — Blood circulation device of CGM MB-1701

SUMMARY:
For Deep Vein Thrombosis (DVT) risk groups, the effect and safety of blood circulation improvement before and after application are evaluated using an investigational device (model name CGM MB-1701).

DETAILED DESCRIPTION:
The investigator applies the test device to the appropriate subjects for a total of 10 days (+1 days) at the institution and nursing hospital, and upon discharge for long-term follow-up investigation, the investigational device is applied at subjects' home according to the subject's consent for about 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women over 19 years of age
2. Subjects who have not been diagnosed with deep vein thrombosis in the lower extremities through the following test results prior to the application of medical devices.

(1) Subjects diagnosed by Doppler ultrasonography as having no blood clots in the femoral vein and the vena poplitea (2) D-dimer negative test result (Even if D-dimer is tested positive, it can be selected through additional tests at the discretion of investigator.)

3. Subjects have 2 or more points of venous thromboembolism (hereinafter referred to as VTE) clinical prediction score (Two-level wells score) at the time of screening.

4. Subjects who fully understand the purpose and procedure of the study and wish to participate in clinical trials with voluntary consent

Exclusion Criteria:

1. Subjects complain of a decrease in the sensation of the lower extremities or is unable to feel the sensation of pain
2. Subjects have inflammation or trauma on the skin that directly touches the device

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Peak Systolic Velocity (PSV) change | 10 days from the baseline
  Compare the PSV change in the right lower extremity femoral vein at 10 days (V4) after application of the test device compared to the baseline (V2).

SECONDARY OUTCOMES:
Peak Systolic Velocity (PSV) change | 5 days from the baseline
  Compare the PSV change in the right lower extremity femoral vein at 5 days (V3) after application of the test device compared to the baseline (V2).
Anteroposterior (AP) diameter | 5 days (V3) and 10 days (V4) from the baseline
  Compare the maximum AP diameter change of the right lower femoral vein at 5 days (V3) and 10 days (V4) after the application of the test device compared to the baseline (V2).
Cross Sectional Area (CSA) | 5 days (V3) and 10 days (V4) from the baseline
  Compare the maximum CSA change of the right lower femoral vein at 5 days (V3) and 10 days (V4) after the application of the test device compare to the baseline (V2).
Leg volume (3D scanner) | 5 days (V3) and 10 days (V4) from the baseline
  Compare the amount of change in leg volume (3D scanner) (left and right) after application at 5 days (V3) and 10 days (V4) compared to the baseline (V2).

CONTACTS AND LOCATIONS:
Overall Officials: Joon-shik Yoon, MD, Principal Investigator — Korea University Guro Hospital
Locations (3):
- South Korea (3):
  - Presbyterian Medical Center, Jeonju
  - Korea University Guro Hospital, Seoul
  - Seoul National University Bundang Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No